CLINICAL TRIAL: NCT00798083
Title: Topical Amitriptyline, Ketamine and Lidocaine in Neuropathic Pain Caused by Radiation Skin Reaction: a Pilot Study
Brief Title: Neuropathic Pain Caused by Radiation Therapy
Acronym: NP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Isabella Uzaraga, British Columbia Cancer Agency - Vancouver Island Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCCA001
Record Dates: First submitted 2008-11-21; First posted 2008-11-25 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Neuropathic Pain Secondary to Radiation Therapy
MeSH Terms: interventions — Amitriptyline; Ketamine; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: topical amitriptyline 2%, ketamine 1%, and lidocaine 5% in pluronic lecitine organogel(AKL in PLO gel) — Subjects will be taught to apply topical 2%amitriptyline, 1% ketamine and 5% lidocaine(AKL) in PLO gel to the sites of maximum neuropathic pain three times per day for up to 2 weeks after completion of radiotherapy.

SUMMARY:
To investigate if topical amitriptyline 2%, ketamine 1%, and lidocaine 5% in pluronic lecitine organogel (AKL in PLO gel) can improve management of neuropathic pain from radiation skin reactions adjunctively or better than standard treatment.

DETAILED DESCRIPTION:
1. Topical amitriptyline and ketamine and topical lidocaine alone have been shown to improve management of neuropathic pain in nonmalignant subjects. Anecdotal experience has shown improvement in use of all three topical drugs combined in radiation skin reactions. There currently is no research evidence for the use of all three compounded interventions. This study aims to target subjects with pain from radiation therapy who are not receiving adequate relief with standard interventions and may be eligible to receive this alternate intervention.
2. Hypothesis:Topical AKL in PLO gel can effectively and safely reduce neuropathic pain experienced by patients with radiotherapy induced skin reactions.
3. Justification: Standard treatment of painful radiation skin reactions such as moist desquamation consists of saline soaks, silver sulfadiazine and oral analgesics. However, sometimes the pain exceeds this standard intervention, patients are sulfa allergic or patients are intolerant to oral analgesics such as opioids. AKL in PLO gel is targeted for neuropathic pain and may be used alternatively to standard interventions. The participation rate will help to further estimate the feasibility of a larger sample size study to look at efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 18 years with ability to provide written informed consent.
* Subjects currently receiving radiation therapy or having completed radiotherapy in less than 4 weeks from study entry, who have developed skin reactions that are painful.
* Radiation skin reaction pain has qualities of burning as scored on UWNPS of 1 or more
* Skin toxicity Assessment Tool showing dry desquamation or worse
* Presence of objective dynamic allodynia and/or pinprick hyperalgesia as assessed by physician
* Subjects show less than 1 point decrease in UWNPS after 2 days of using standard intervention.
* Subjects are allergic or intolerant to standard intervention.
* Subjects must be available by telephone 2 and 6 weeks after RT treatment is completed.

Exclusion Criteria:

* Allergy to amitriptyline, ketamine or lidocaine
* Untreated severe major depression
* Ongoing use of monoamine oxidase inhibitor
* Pain from another source as severe or greater than the pain under study
* Evidence of another type of neuropathic pain not included in this study.
* Normal cognitive and communicative ability as judged by clinical assessment and ability to complete self-report questionnaires
* Not pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will to use the validated University of Washington Neuropathic Pain Scale (UWNPS) on all radiation skin reaction subjects requiring standard intervention. | University of Washington Neuropathic Pain scale will be conducted at the time of assessment, every 2-5 days while on radiotherapy, week 2 and 6 weeks post radiotherapy.

SECONDARY OUTCOMES:
Skin Toxicity Assessment Tool (STAT) | Presence of dry desquamation or worse on STAT at baseline assessment, complete STAT 30 minutes post application of cream, every 2-5 days while on radiotherapy, week 2 and 6 weeks after completing radiation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Uzaraga, MD, Principal Investigator — BC Cancer Agency - Vancouver Island Centre
Locations (1):
- BC Cancer Agency Vancouver Island BCCA, Victoria, British Columbia, Canada